CLINICAL TRIAL: NCT02771093
Title: An Exploratory Study to Evaluate the Effects of Trelagliptin and Alogliptin by CGM on Glucose Variability for One Week in Patients With Type 2 Diabetes Mellitus
Brief Title: An Exploratory Study of the Effects of Trelagliptin and Alogliptin on Glucose Variability in Patients With Type 2 Diabetes Mellitus
Acronym: TRACK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Trelagliptin-4001; U1111-1182-4062 (Other: UTN); JapicCTI-163250 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2016-05-11; First posted 2016-05-12 (Estimated); Results first posted 2018-12-10 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2, Diabetes, Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — trelagliptin; alogliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trelagliptin 100 mg group (Experimental): Trelagliptin 100 mg once weekly taken orally before breakfast
  Interventions: Drug: Trelagliptin
- Alogliptin 25 mg group (Experimental): Alogliptin 25 mg once daily taken orally before breakfast
  Interventions: Drug: Alogliptin

INTERVENTIONS:
Drug: Trelagliptin — Trelagliptin 100 mg tablet
  Arms: Trelagliptin 100 mg group
Drug: Alogliptin — Alogliptin 25 mg tablet
  Arms: Alogliptin 25 mg group

SUMMARY:
This is a multi-center, randomized, open-label, parallel-group comparative, exploratory study to evaluate the effect of trelagliptin administered at a dose of 100 mg once weekly or alogliptin administered at a dose of 25 mg once daily for 4 weeks on glycemic variation in patients with type 2 diabetes mellitus using continuous glucose monitoring (CGM).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of trelagliptin administered orally at a dose of 100 mg once weekly or alogliptin administered orally at a dose of 25 mg once daily for 4 weeks on glycemic variation in an exploratory manner as a primary objective and to evaluate the effect of difference method of administration of Dipeptidyl-peptidase (DPP)-4 on glycemic variation as secondary objective.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who, in the opinion of the principal investigator or the investigator, are capable of understanding the content of the clinical research and complying with the research protocol requirements.
2. Participants who are able to sign and date the informed consent form and information sheet prior to the start of study procedures.
3. Participants diagnosed with type 2 diabetes mellitus.
4. Participants with a glycated hemoglobin (HbA1c) [National Glycohemoglobin Standardization Program (NGSP value)] value ≥ 6.5% and < 8.5% at the start of the observation period (Day -2).
5. Participants who experience a ≤ ±1.0% change in HbA1c (NGSP value) at the start of the observation period (Day -2) as compared with an HbA1c value obtained during the preceding 6 weeks.
6. Participants receiving stable dietetic therapy and exercise therapy (if performed) for ≥ 4 weeks before the start of the observation period.
7. Participants, who in the opinion of the principal investigator or the investigator, does not have to change (including discontinuation or interruption) 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) reductase inhibitors or add new HMG-CoA reductase inhibitors during treatment period.
8. Men or women aged 20 years or older at the time of informed consent.

Exclusion Criteria:

1. Participants who received anti-diabetic medications within 4 weeks prior to the start of the observation period.
2. Participants who have changed (including discontinuation or interruption) HMG-CoA reductase inhibitors or received new HMG-CoA reductase inhibitors ≤ 4 weeks before the start of the observation period.
3. Participants with clinically evident hepatic dysfunction (e.g., aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 2.5-fold the upper limit of normal at the start of the observation period [Day -2]).
4. Participants with moderate renal dysfunction, severe renal dysfunction or renal failure (e.g., creatinine clearance < 50 mL/min or serum creatinine > 1.4 mg/dL in men or > 1.2 mg/dL in women [equivalent to the creatinine clearance for persons aged 60 years with a body weight of 65 kg] at the start of the observation period [Day -2]).
5. Participants with severe heart disease, cerebrovascular disorder, or severe pancreatic, hematologic or other diseases.
6. Participants with a history of gastric or small intestinal resection.
7. Participants with proliferative diabetic retinopathy.
8. Participants warranting insulin therapy for glycemic control (e.g., participants with severe ketosis, diabetic coma or precoma, type 1 diabetes mellitus, severe infection, perioperative participants, or serious trauma).
9. Participants with a history of hypersensitivity or allergy to DPP-4 inhibitors.
10. Participants who experience an allergic reaction to metal during CGM at the start of the observation period (Day -2).
11. Participants with any malignant tumors.
12. Habitual drinkers whose average daily alcohol consumption is > 100 mL.
13. Participants who have any contraindications for the study drug or are taking any contraindicated concomitant drugs listed in the package insert.
14. Participants anticipated to require any prohibited concomitant medications during the study period.
15. Participants who are day and night lifestyle reversal.
16. Participants participating in any other clinical studies at the time of informed consent for this study.
17. Pregnant women, nursing mothers, women who are possible pregnant, or women who plan to become pregnant.
18. Other participants who are considered inappropriate for participation in this study in the opinion of the principal investigator or investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-09-08 (Actual); Primary Completion 2017-04-27 (Actual); Study Completion 2017-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Naka, Ibaragi, Japan

REFERENCES:
- [Derived] Nishimura R, Osonoi T, Koike Y, Miyata K, Shimasaki Y. A Randomized Pilot Study of the Effect of Trelagliptin and Alogliptin on Glycemic Variability in Patients with Type 2 Diabetes. Adv Ther. 2019 Nov;36(11):3096-3109. doi: 10.1007/s12325-019-01097-z. Epub 2019 Sep 27. PMID 31562608

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in Japan, from 08 September 2016 to 27 April 2017.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus were enrolled in 1 of 2 (the trelagliptin 100 mg group or the alogliptin 25 mg group) treatment groups.
Groups:
- Trelagliptin 100 mg: Trelagliptin 100 mg group; Trelagliptin 100 mg once weekly taken orally before breakfast.
- Alogliptin 25 mg: Alogliptin 25 mg group; Alogliptin 25 mg once daily taken orally before breakfast.
Period: Overall Study
Arm/Group | Trelagliptin 100 mg | Alogliptin 25 mg
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS); FAS was defined as participants who were randomized and received at least one dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trelagliptin 100 mg | Alogliptin 25 mg | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (10.14) | 62.7 (7.64) | 62.7 (8.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 7 | 10 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Japan | 13 | 14 | 27
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 160.9 (10.40) | 164.4 (7.17) | 162.7 (8.87)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 66.45 (14.107) | 64.15 (9.585) | 65.26 (11.796)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: (kg/m^2)] — Body Mass Index = weight (kg)/[height (m)^2]
  (kg/m^2) | 25.45 (2.948) | 23.65 (2.404) | 24.52 (2.783)
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 8 | 7 | 15
  Current Smoker | 3 | 3 | 6
  Ex-Smoker | 2 | 4 | 6
Alcohol Classification [Count of Participants; unit: Participants] — Participants who answered Yes or No for a question "Drink Alcohol Almost Every Day?" were reported.
  Participants
    Yes | 1 | 2 | 3
    No | 12 | 12 | 24
Duration of Diabetes Mellitus [Mean (Standard Deviation); unit: years] — Mean duration between start of study and first time of diagnosis of type 2 diabetes mellitus was reported.
  years | 5.62 (4.471) | 6.15 (4.679) | 5.89 (4.500)
Glycated hemoglobin A1c (HbA1c) [National Glycohemoglobin Standardization Program (NGSP)] [Mean (Standard Deviation); unit: percent] | 7.29 (0.616) | 7.19 (0.339) | 7.24 (0.485)
Mean Amplitude Glycemic Excursions (MAGE) [Mean (Standard Deviation); unit: millgrams per deciliter (mg/dL)] — MAGE is used for a measurement of the degree of glucose level fluctuations, and is the average difference of blood glucose levels exceeds 1 standard deviation (SD) of the average 24-hours blood glucose levels. MAGE was calculated from the data of blood glucose levels every day during continuous glucose monitoring (CGM) in the observation and treatment periods. Population: The number analyzed is the number of participants with data available for analysis.
  millgrams per deciliter (mg/dL)
    number analyzed (Participants) | 13 | 13 | 26
    (all) | 98.02 (44.191) | 114.91 (38.454) | 106.47 (41.488)
Mean 24-hour Blood Glucose [Mean (Standard Deviation); unit: mg/dL] | 145.65 (17.570) | 161.01 (18.349) | 153.62 (19.287)
Area Under the Plasma Concentration-time Curve (AUC) of blood glucose [Mean (Standard Deviation); unit: mg*min/dL] | 41947.9 (5058.50) | 46372.7 (5282.47) | 44242.3 (5553.22)
Fasting Insulin [Mean (Standard Deviation); unit: uU/mL] | 9.42 (4.177) | 8.79 (4.395) | 9.09 (4.221)
Fasting Blood Glucose [Mean (Standard Deviation); unit: mg/dL] | 144.0 (17.57) | 145.5 (19.15) | 144.8 (18.06)

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline in the Standard Deviation (SD) of 24-hour Blood Glucose Values
Description: Changes in the SD of 24-hour blood glucose values (mg/dL) for each 7-day period between Week 3 and Week 4 (between Day 2 on Week 3 [Day 22] and Day 8 on Week 3 [Day 28]) of the treatment period, calculated from the value at the start of the observation period.
Time Frame: Baseline, up to 28 days
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Trelagliptin 100 mg | Alogliptin 25 mg
Number analyzed (Participants) | 13 | 14
mg/dL
  Day(D) 2 Week(W) 3 | -7.51 [-17.10 to 2.08] | -13.04 [-20.84 to -5.23]
  D3W3 | -11.76 [-21.12 to -2.40] | -15.24 [-21.87 to -8.61]
  D4W3 | -11.71 [-21.84 to -1.58] | -12.91 [-18.55 to -7.26]
  D5W3 | -9.89 [-19.83 to 0.05] | -13.28 [-21.28 to -5.27]
  D6W3 | -12.75 [-22.01 to -3.49] | -11.94 [-20.58 to -3.29]
  D7W3 | -9.50 [-18.58 to -0.42] | -10.90 [-20.00 to -1.80]
  D8W3 | -7.35 [-15.13 to 0.44] | -11.63 [-18.67 to -4.59]

2. Secondary Outcome: Change From Baseline in AUC for Blood Glucose When Specific Blood Glucose Levels (180 mg/dL) Are Observed During the 3 Hour Time Period After Breakfast, Lunch and Evening Meal
Description: Change from baseline in AUC for blood glucose when specific blood glucose levels (180 mg/dL) were observed during the 3 hour time period after breakfast, lunch and evening meal at each time points was calculated.
Time Frame: Baseline, up to 28 days
Population: Full analysis set (FAS); FAS was defined as participants who were randomized and received at least one dose of the study drug. The number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Mean (95% Confidence Interval); unit: mg·min/dL
Arm/Group | Trelagliptin 100 mg | Alogliptin 25 mg
Number analyzed (Participants) | 13 | 14
mg·min/dL
  D2W3 after breakfast | -90.7 [-559.9 to 378.5] | -660.1 [-1128.5 to -191.6]
  D3W3 after breakfast | -241.2 [-841.3 to 359.0] | -592.9 [-1016.9 to -169.0]
  D4W3 after breakfast: number analyzed (Participants) | 5 | 10
  D4W3 after breakfast | -632.2 [-1357.8 to 93.4] | -375.6 [-827.9 to 76.7]
  D5W3 after breakfast: number analyzed (Participants) | 11 | 8
  D5W3 after breakfast | 36.5 [-418.1 to 491.2] | -776.3 [-1602.1 to 49.6]
  D6W3 after breakfast: number analyzed (Participants) | 13 | 11
  D6W3 after breakfast | -272.2 [-673.5 to 129.0] | -556.5 [-1099.4 to -13.7]
  D7W3 after breakfast | -264.2 [-803.3 to 274.8] | -578.2 [-1000.6 to -155.8]
  D8W3 after breakfast | -214.8 [-639.5 to 209.8] | -603.6 [-1005.5 to -201.8]
  D2W3 after lunch | -300.3 [-924.2 to 323.6] | -626.6 [-1126.4 to -126.7]
  D3W3 after lunch | -383.8 [-936.3 to 168.7] | -521.1 [-1048.5 to 6.3]
  D4W3 after lunch | -307.0 [-878.0 to 264.0] | -404.1 [-890.6 to 82.3]
  D5W3 after lunch | -430.4 [-989.5 to 128.7] | -589.9 [-1093.1 to -86.6]
  D6W3 after lunch | -353.5 [-859.1 to 152.2] | -354.6 [-979.3 to 270.1]
  D7W3 after lunch | -184.2 [-697.4 to 329.1] | -293.6 [-923.6 to 336.3]
  D8W3 after lunch | -234.0 [-767.7 to 299.7] | -546.4 [-1085.4 to -7.4]
  D2W3 after evening meal | -507.6 [-1077.9 to 62.7] | -375.9 [-841.4 to 89.7]
  D3W3 after evening meal | -592.4 [-1198.5 to 13.8] | -484.4 [-1022.2 to 53.5]
  D4W3 after evening meal | -662.4 [-1251.3 to -73.4] | -597.2 [-1070.4 to -124.0]
  D5W3 after evening meal: number analyzed (Participants) | 13 | 13
  D5W3 after evening meal | -641.9 [-1202.6 to -81.2] | -427.8 [-1024.2 to 168.5]
  D6W3 after evening meal | -598.8 [-1183.3 to -14.4] | -552.4 [-1101.3 to -3.5]
  D7W3 after evening meal | -612.6 [-1195.8 to -29.4] | -374.5 [-1024.4 to 275.4]
  D8W3 after evening meal | -555.4 [-1128.7 to 17.9] | -346.5 [-895.1 to 202.1]

3. Secondary Outcome: Change From Baseline in AUC for Blood Glucose When Specific Blood Glucose Levels (110 mg/dL) Are Observed During the 3 Hour Time Period After Breakfast, Lunch and Evening Meal
Description: Change from baseline in AUC for blood glucose when specific blood glucose levels (110 mg/dL) were observed during the 3 hour time period after breakfast, lunch and evening meal at each time points was calculated.
Time Frame: Baseline, up to 28 days
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg·min/dL
Arm/Group | Trelagliptin 100 mg | Alogliptin 25 mg
Number analyzed (Participants) | 13 | 14
mg·min/dL
  D2W3 after breakfast | -203.7 [-857.5 to 450.1] | -1052.7 [-1596.7 to -508.7]
  D3W3 after breakfast | -662.6 [-1590.9 to 265.7] | -1030.9 [-1538.5 to -523.4]
  D4W3 after breakfast: number analyzed (Participants) | 5 | 10
  D4W3 after breakfast | -1024.6 [-2341.3 to 292.1] | -958.9 [-1723.4 to -194.4]
  D5W3 after breakfast: number analyzed (Participants) | 11 | 8
  D5W3 after breakfast | -97.2 [-808.5 to 614.2] | -1319.8 [-2358.8 to -280.7]
  D6W3 after breakfast: number analyzed (Participants) | 13 | 11
  D6W3 after breakfast | -696.1 [-1333.9 to -58.3] | -832.5 [-1606.6 to -58.4]
  D7W3 after breakfast | -573.8 [-1309.2 to 161.5] | -966.3 [-1566.5 to -366.0]
  D8W3 after breakfast | -399.0 [-1034.8 to 236.8] | -1024.8 [-1550.4 to -499.2]
  D2W3 after lunch | -669.0 [-1648.8 to 310.8] | -1131.4 [-1738.4 to -524.5]
  D3W3 after lunch | -500.1 [-1269.9 to 269.7] | -941.9 [-1716.5 to -167.4]
  D4W3 after lunch | -468.2 [-1272.1 to 335.6] | -701.1 [-1330.5 to -71.8]
  D5W3 after lunch | -793.5 [-1682.3 to 95.2] | -1065.4 [-1736.4 to -394.3]
  D6W3 after lunch | -798.5 [-1554.0 to -43.1] | -534.4 [-1276.7 to 207.8]
  D7W3 after lunch | -320.4 [-1078.0 to 437.2] | -488.7 [-1297.0 to 319.6]
  D8W3 after lunch | -521.3 [-1377.2 to 334.6] | -923.5 [-1700.5 to -146.5]
  D2W3 after evening meal | -1079.4 [-1793.3 to -365.4] | -800.5 [-1381.4 to -219.6]
  D3W3 after evening meal | -1273.0 [-2148.7 to -397.3] | -1023.6 [-1676.2 to -371.1]
  D4W3 after evening meal | -1359.6 [-2101.2 to -618.0] | -1228.5 [-1793.6 to -663.4]
  D5W3 after evening meal: number analyzed (Participants) | 13 | 13
  D5W3 after evening meal | -1351.4 [-2063.7 to -639.0] | -756.1 [-1532.4 to 20.3]
  D6W3 after evening meal | -1199.9 [-1847.4 to -552.4] | -1144.2 [-1786.6 to -501.9]
  D7W3 after evening meal | -884.2 [-1659.0 to -109.3] | -669.9 [-1432.0 to 92.1]
  D8W3 after evening meal | -1142.0 [-2041.2 to -242.8] | -577.0 [-1218.8 to 64.8]

4. Secondary Outcome: Change From Baseline in AUC for Blood Glucose When Specific Blood Glucose Levels (140 mg/dL) Are Observed During the 3 Hour Time Period After Breakfast, Lunch and Evening Meal
Description: Change from baseline in AUC for blood glucose when specific blood glucose levels (140 mg/dL) were observed during the 3 hour time period after breakfast, lunch and evening meal at each time points was calculated.
Time Frame: Baseline, up to 28 days
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg·min/dL
Arm/Group | Trelagliptin 100 mg | Alogliptin 25 mg
Number analyzed (Participants) | 13 | 14
mg·min/dL
  D2W3 after breakfast | -218.5 [-811.5 to 374.4] | -981.2 [-1502.5 to -459.9]
  D3W3 after breakfast | -510.2 [-1377.6 to 357.2] | -926.1 [-1418.1 to -434.2]
  D4W3 after breakfast: number analyzed (Participants) | 5 | 10
  D4W3 after breakfast | -886.4 [-1860.8 to 88.0] | -801.6 [-1487.3 to -115.9]
  D5W3 after breakfast: number analyzed (Participants) | 11 | 8
  D5W3 after breakfast | -21.3 [-672.0 to 629.4] | -1178.0 [-2185.7 to -170.3]
  D6W3 after breakfast: number analyzed (Participants) | 13 | 11
  D6W3 after breakfast | -559.8 [-1140.7 to 21.0] | -791.8 [-1517.5 to -66.2]
  D7W3 after breakfast | -457.4 [-1154.7 to 239.9] | -910.1 [-1492.1 to -328.1]
  D8W3 after breakfast | -348.5 [-942.4 to 245.5] | -951.6 [-1450.0 to -453.1]
  D2W3 after lunch | -588.5 [-1518.0 to 340.9] | -1079.1 [-1649.8 to -508.5]
  D3W3 after lunch | -489.7 [-1242.6 to 263.2] | -845.4 [-1573.8 to -116.9]
  D4W3 after lunch | -429.3 [-1195.4 to 336.8] | -648.1 [-1253.9 to -42.3]
  D5W3 after lunch | -725.5 [-1549.9 to 99.0] | -970.0 [-1560.0 to -380.0]
  D6W3 after lunch | -707.9 [-1383.0 to -32.9] | -517.0 [-1245.9 to 211.9]
  D7W3 after lunch | -294.9 [-1014.3 to 424.4] | -458.3 [-1237.2 to 320.6]
  D8W3 after lunch | -474.7 [-1254.4 to 305.0] | -867.4 [-1598.8 to -135.9]
  D2W3 after evening meal | -950.8 [-1638.1 to -263.4] | -637.6 [-1184.9 to -90.2]
  D3W3 after evening meal | -1077.3 [-1902.8 to -251.8] | -862.0 [-1508.7 to -215.3]
  D4W3 after evening meal | -1147.1 [-1874.5 to -419.6] | -1016.8 [-1565.1 to -468.4]
  D5W3 after evening meal: number analyzed (Participants) | 13 | 13
  D5W3 after evening meal | -1147.5 [-1841.6 to -453.3] | -613.7 [-1369.9 to 142.5]
  D6W3 after evening meal | -1030.6 [-1668.4 to -392.8] | -966.4 [-1594.0 to -338.7]
  D7W3 after evening meal | -822.3 [-1561.4 to -83.2] | -586.4 [-1346.1 to 173.4]
  D8W3 after evening meal | -964.8 [-1812.4 to -117.1] | -535.0 [-1170.4 to 100.4]

5. Secondary Outcome: Change From Baseline in AUC for Blood Glucose When Specific Blood Glucose Levels (160 mg/dL) Are Observed During the 3 Hour Time Period After Breakfast, Lunch and Evening Meal
Description: Change from baseline in AUC for blood glucose when specific blood glucose levels (160 mg/dL) were observed during the 3 hour time period after breakfast, lunch and evening meal at each time points was calculated.
Time Frame: Baseline, up to 28 days
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg·min/dL
Arm/Group | Trelagliptin 100 mg | Alogliptin 25 mg
Number analyzed (Participants) | 13 | 14
mg·min/dL
  D2W3 after breakfast | -164.5 [-704.0 to 374.9] | -829.2 [-1327.2 to -331.2]
  D3W3 after breakfast | -377.8 [-1142.0 to 386.4] | -770.4 [-1225.2 to -315.5]
  D4W3 after breakfast: number analyzed (Participants) | 5 | 10
  D4W3 after breakfast | -759.4 [-1568.6 to 49.8] | -609.9 [-1198.1 to -21.7]
  D5W3 after breakfast: number analyzed (Participants) | 11 | 8
  D5W3 after breakfast | 25.6 [-546.2 to 597.5] | -981.3 [-1918.9 to -43.6]
  D6W3 after breakfast: number analyzed (Participants) | 13 | 11
  D6W3 after breakfast | -405.5 [-912.4 to 101.5] | -696.8 [-1340.7 to -53.0]
  D7W3 after breakfast | -356.6 [-1001.3 to 288.0] | -760.4 [-1278.1 to -242.6]
  D8W3 after breakfast | -273.4 [-787.3 to 240.5] | -806.3 [-1259.2 to -353.4]
  D2W3 after lunch | -448.1 [-1249.4 to 353.2] | -890.4 [-1433.1 to -347.7]
  D3W3 after lunch | -462.2 [-1122.9 to 198.6] | -705.5 [-1346.4 to -64.6]
  D4W3 after lunch | -389.7 [-1066.5 to 287.1] | -552.5 [-1109.1 to 4.1]
  D5W3 after lunch | -579.4 [-1289.4 to 130.6] | -811.9 [-1359.0 to -264.9]
  D6W3 after lunch | -534.1 [-1126.5 to 58.4] | -469.7 [-1161.5 to 222.1]
  D7W3 after lunch | -249.9 [-884.3 to 384.4] | -384.6 [-1104.5 to 335.3]
  D8W3 after lunch | -350.8 [-1014.3 to 312.8] | -730.1 [-1384.0 to -76.2]
  D2W3 after evening meal | -730.5 [-1380.6 to -80.3] | -507.4 [-1016.6 to 1.9]
  D3W3 after evening meal | -825.2 [-1545.9 to -104.4] | -671.1 [-1284.7 to -57.5]
  D4W3 after evening meal | -914.5 [-1611.8 to -217.2] | -808.9 [-1337.7 to -280.2]
  D5W3 after evening meal: number analyzed (Participants) | 13 | 13
  D5W3 after evening meal | -887.5 [-1532.6 to -242.5] | -508.3 [-1195.0 to 178.4]
  D6W3 after evening meal | -809.5 [-1436.6 to -182.4] | -759.6 [-1361.2 to -157.9]
  D7W3 after evening meal | -742.3 [-1403.7 to -81.0] | -504.1 [-1235.0 to 226.7]
  D8W3 after evening meal | -763.4 [-1480.9 to -45.8] | -460.2 [-1059.2 to 138.8]

6. Secondary Outcome: Change From Baseline in AUC for Blood Glucose During Periods When Blood Glucose Levels Reached 140 mg/dL (Hyperglycemia)
Description: Change from baseline in AUC for blood glucose during periods when blood glucose levels reached 140 mg/dL at each time points was calculated.
Time Frame: Baseline, up to 28 days
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: mg·min/dL
Arm/Group | Trelagliptin 100 mg | Alogliptin 25 mg
Number analyzed (Participants) | 13 | 14
mg·min/dL
  D2W3 | -1935.9 [-4619.7 to 747.9] | -4021.4 [-5867.0 to -2175.7]
  D3W3 | -2001.2 [-4861.6 to 859.3] | -3378.3 [-6054.9 to -701.7]
  D4W3 | -2978.2 [-5095.6 to -860.8] | -4119.9 [-5855.8 to -2384.1]
  D5W3 | -2981.5 [-5010.4 to -952.5] | -4230.4 [-6524.2 to -1936.7]
  D6W3 | -2550.5 [-4308.5 to -792.4] | -3840.0 [-6136.0 to -1544.0]
  D7W3 | -1946.5 [-3589.5 to -303.5] | -3566.4 [-5763.1 to -1369.6]
  D8W3 | -2043.5 [-4237.3 to 150.4] | -3667.1 [-5489.4 to -1844.7]

7. Secondary Outcome: Change From Baseline in AUC for Blood Glucose During Periods When Blood Glucose Levels Reached 160 mg/dL (Hyperglycemia)
Description: Change from baseline in AUC for blood glucose during periods when blood glucose levels reached 160 mg/dL at each time points was calculated.
Time Frame: Baseline, up to 28 days
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: mg·min/dL
Arm/Group | Trelagliptin 100 mg | Alogliptin 25 mg
Number analyzed (Participants) | 13 | 14
mg·min/dL
  D2W3 | -1458.0 [-3556.4 to 640.4] | -3075.8 [-4672.5 to -1479.1]
  D3W3 | -1702.0 [-3893.0 to 489.0] | -2767.3 [-4792.8 to -741.8]
  D4W3 | -2335.8 [-4011.2 to -660.3] | -3273.0 [-4820.1 to -1725.9]
  D5W3 | -2171.8 [-3923.9 to -419.8] | -3384.5 [-5073.8 to -1695.2]
  D6W3 | -2031.0 [-3588.9 to -473.1] | -2990.8 [-4843.0 to -1138.6]
  D7W3 | -1636.5 [-3081.2 to -191.9] | -2768.9 [-4705.6 to -832.1]
  D8W3 | -1603.9 [-3357.3 to 149.5] | -2818.8 [-4272.4 to -1365.2]

8. Secondary Outcome: Change From Baseline in AUC for Blood Glucose During Periods When Blood Glucose Levels Reached 180 mg/dL (Hyperglycemia)
Description: Change from baseline in AUC for blood glucose during periods when blood glucose levels reached 180 mg/dL at each time points was calculated.
Time Frame: Baseline, up to 28 days
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: mg·min/dL
Arm/Group | Trelagliptin 100 mg | Alogliptin 25 mg
Number analyzed (Participants) | 13 | 14
mg·min/dL
  D2W3 | -989.9 [-2508.3 to 528.4] | -2247.9 [-3524.3 to -971.6]
  D3W3 | -1332.7 [-2948.0 to 282.6] | -2086.7 [-3524.9 to -648.5]
  D4W3 | -1685.1 [-3054.1 to -316.0] | -2352.2 [-3639.5 to -1065.0]
  D5W3 | -1486.5 [-2877.5 to -95.5] | -2492.3 [-3775.9 to -1208.6]
  D6W3 | -1449.4 [-2803.7 to -95.0] | -2109.1 [-3559.9 to -658.2]
  D7W3 | -1264.2 [-2516.7 to -11.8] | -1976.3 [-3590.5 to -362.1]
  D8W3 | -1166.8 [-2536.5 to 202.8] | -2009.8 [-3116.4 to -903.2]

9. Secondary Outcome: Change From Baseline in Time During Periods When Blood Glucose Levels Reached 140 mg/dL (Hyperglycemia)
Description: Change from baseline in cumulative time during periods when blood glucose levels reached 140 mg/dL at each time points was calculated.
Time Frame: Baseline, up to 28 days
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: min
Arm/Group | Trelagliptin 100 mg | Alogliptin 25 mg
Number analyzed (Participants) | 13 | 14
min
  D2W3 | -116.9 [-321.9 to 88.1] | -212.5 [-326.5 to -98.5]
  D3W3 | -105.0 [-318.1 to 108.1] | -147.1 [-353.5 to 59.2]
  D4W3 | -163.8 [-338.4 to 10.8] | -166.1 [-312.4 to -19.8]
  D5W3 | -192.3 [-363.7 to -20.9] | -163.2 [-376.8 to 50.4]
  D6W3 | -114.2 [-300.0 to 71.5] | -193.2 [-370.9 to -15.6]
  D7W3 | -96.9 [-243.3 to 49.5] | -182.1 [-325.5 to -38.8]
  D8W3 | -133.8 [-328.2 to 60.5] | -198.6 [-348.0 to -49.2]

10. Secondary Outcome: Change From Baseline in Time During Periods When Blood Glucose Levels Reached 160 mg/dL (Hyperglycemia)
Description: Change from baseline in cumulative time during periods when blood glucose levels reached 160 mg/dL at each time points was calculated.
Time Frame: Baseline, up to 28 days
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: min
Arm/Group | Trelagliptin 100 mg | Alogliptin 25 mg
Number analyzed (Participants) | 13 | 14
min
  D2W3 | -134.2 [-315.6 to 47.1] | -229.3 [-329.7 to -128.9]
  D3W3 | -75.0 [-291.9 to 141.9] | -173.2 [-356.0 to 9.6]
  D4W3 | -167.7 [-322.8 to -12.6] | -234.3 [-331.5 to -137.0]
  D5W3 | -200.0 [-323.0 to -77.0] | -236.8 [-389.3 to -84.2]
  D6W3 | -153.1 [-287.4 to -18.7] | -232.9 [-361.4 to -104.3]
  D7W3 | -93.5 [-209.1 to 22.1] | -213.2 [-328.9 to -97.5]
  D8W3 | -115.0 [-255.6 to 25.6] | -225.4 [-339.3 to -111.4]

11. Secondary Outcome: Change From Baseline in Time During Periods When Blood Glucose Levels Reached 180 mg/dL (Hyperglycemia)
Description: Change from baseline in cumulative time during periods when blood glucose levels reached 180 mg/dL at each time points was calculated.
Time Frame: Baseline, up to 28 days
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: min
Arm/Group | Trelagliptin 100 mg | Alogliptin 25 mg
Number analyzed (Participants) | 13 | 14
min
  D2W3 | -91.2 [-255.3 to 73.0] | -210.7 [-315.9 to -105.6]
  D3W3 | -117.3 [-271.7 to 37.1] | -167.1 [-324.6 to -9.7]
  D4W3 | -167.3 [-262.0 to -72.6] | -236.4 [-339.0 to -133.8]
  D5W3 | -153.1 [-273.6 to -32.6] | -225.4 [-341.4 to -109.4]
  D6W3 | -137.7 [-234.0 to -41.4] | -216.8 [-336.1 to -97.5]
  D7W3 | -94.2 [-185.2 to -3.2] | -194.3 [-308.5 to -80.1]
  D8W3 | -105.0 [-232.7 to 22.7] | -193.2 [-290.5 to -96.0]

12. Secondary Outcome: Change From Baseline in AUC for Blood Glucose During Periods When Blood Glucose Levels is Less Than 70 mg/dL (Hypoglycemia)
Description: Change from baseline in AUC for blood glucose during periods when blood glucose levels was less than 70 mg/dL at each time points was calculated.
Time Frame: Baseline, up to 28 days
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: mg·min/dL
Arm/Group | Trelagliptin 100 mg | Alogliptin 25 mg
Number analyzed (Participants) | 13 | 14
mg·min/dL
  D2W3 | -31.2 [-105.8 to 43.3] | 0.4 [-0.4 to 1.1]
  D3W3 | -43.0 [-136.3 to 50.3] | 0.0 [0.0 to 0.0]
  D4W3 | -42.3 [-135.8 to 51.2] | 13.4 [-14.0 to 40.8]
  D5W3 | -30.5 [-129.9 to 68.8] | 26.9 [-8.9 to 62.6]
  D6W3 | -39.8 [-134.0 to 54.3] | 0.0 [0.0 to 0.0]
  D7W3 | -43.0 [-136.3 to 50.3] | 0.0 [0.0 to 0.0]
  D8W3 | -43.0 [-136.3 to 50.3] | 0.0 [0.0 to 0.0]

13. Secondary Outcome: Change From Baseline in Peak Postprandial Glucose Levels During the 3 Hour Time Period After Breakfast, Lunch and Evening Meal
Description: Change from baseline in peak postprandial glucose levels during the 3 hour time period after breakfast, lunch and evening meal at each time points was calculated.
Time Frame: Baseline, up to 28 days
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Trelagliptin 100 mg | Alogliptin 25 mg
Number analyzed (Participants) | 13 | 14
mg/dL
  D2W3 after breakfast | -11.3 [-45.9 to 23.3] | -35.6 [-55.1 to -16.0]
  D3W3 after breakfast | -35.4 [-70.1 to -0.6] | -29.1 [-50.0 to -8.1]
  D4W3 after breakfast: number analyzed (Participants) | 5 | 10
  D4W3 after breakfast | -39.4 [-86.6 to 7.8] | -29.0 [-54.3 to -3.7]
  D5W3 after breakfast: number analyzed (Participants) | 11 | 8
  D5W3 after breakfast | -4.9 [-34.0 to 24.2] | -41.1 [-70.3 to -11.9]
  D6W3 after breakfast: number analyzed (Participants) | 13 | 11
  D6W3 after breakfast | -28.6 [-51.9 to -5.4] | -24.2 [-50.1 to 1.7]
  D7W3 after breakfast | -23.7 [-56.7 to 9.3] | -29.6 [-51.6 to -7.5]
  D8W3 after breakfast | -16.6 [-44.6 to 11.4] | -31.4 [-55.6 to -7.2]
  D2W3 after lunch | -26.9 [-66.1 to 12.2] | -40.8 [-63.8 to -17.8]
  D3W3 after lunch | -25.9 [-55.8 to 3.9] | -35.1 [-63.6 to -6.7]
  D4W3 after lunch | -21.9 [-51.5 to 7.7] | -16.6 [-42.6 to 9.3]
  D5W3 after lunch | -34.8 [-67.4 to -2.2] | -41.6 [-68.3 to -14.9]
  D6W3 after lunch | -32.7 [-63.0 to -2.4] | -18.7 [-50.8 to 13.4]
  D7W3 after lunch | -11.5 [-44.7 to 21.8] | -18.1 [-48.6 to 12.3]
  D8W3 after lunch | -17.7 [-49.2 to 13.8] | -33.6 [-63.7 to -3.6]
  D2W3 after evening meal | -40.6 [-68.4 to -12.9] | -21.3 [-44.3 to 1.8]
  D3W3 after evening meal | -44.5 [-82.2 to -6.7] | -21.6 [-45.0 to 1.7]
  D4W3 after evening meal | -45.8 [-78.6 to -13.0] | -32.7 [-50.8 to -14.6]
  D5W3 after evening meal: number analyzed (Participants) | 13 | 13
  D5W3 after evening meal | -40.6 [-69.3 to -12.0] | -15.6 [-43.2 to 12.0]
  D6W3 after evening meal | -41.5 [-68.0 to -15.0] | -33.8 [-57.2 to -10.4]
  D7W3 after evening meal | -32.3 [-59.1 to -5.5] | -13.9 [-42.8 to 15.0]
  D8W3 after evening meal | -42.2 [-73.3 to -11.2] | -15.9 [-35.7 to 3.8]

14. Secondary Outcome: Change From Baseline in Maximum Variation of Blood Glucose Levels Between Before and After Breakfast, Lunch, and Evening Meal
Description: Change from baseline in maximum variation of glucose levels between before and after breakfast, lunch and evening meal at each time points was calculated.
Time Frame: Baseline, up to 28 days
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Trelagliptin 100 mg | Alogliptin 25 mg
Number analyzed (Participants) | 13 | 14
mg/dL
  D2W3 between before/after breakfast | -13.9 [-51.7 to 23.8] | -28.9 [-54.0 to -3.7]
  D3W3 between before/after breakfast | -47.4 [-77.3 to -17.5] | -35.4 [-57.6 to -13.1]
  D4W3 between before/after breakfast: number analyzed (Participants) | 5 | 10
  D4W3 between before/after breakfast | -41.2 [-77.7 to -4.7] | -42.1 [-70.2 to -14.0]
  D5W3 between before/after breakfast: number analyzed (Participants) | 11 | 8
  D5W3 between before/after breakfast | -7.0 [-25.1 to 11.1] | -25.5 [-55.6 to 4.6]
  D6W3 between before/after breakfast: number analyzed (Participants) | 13 | 11
  D6W3 between before/after breakfast | -38.6 [-65.9 to -11.4] | -29.8 [-62.3 to 2.7]
  D7W3 between before/after breakfast | -36.4 [-67.2 to -5.6] | -33.3 [-58.2 to -8.4]
  D8W3 between before/after breakfast | -36.2 [-61.0 to -11.3] | -34.5 [-58.8 to -10.2]
  D2W3 between before/after lunch | -30.2 [-66.2 to 5.7] | -35.5 [-64.4 to -6.6]
  D3W3 between before/after lunch | -34.5 [-68.9 to -0.1] | -29.5 [-61.3 to 2.3]
  D4W3 between before/after lunch | -23.8 [-59.2 to 11.5] | -6.2 [-39.1 to 26.6]
  D5W3 between before/after lunch | -34.8 [-73.8 to 4.2] | -31.2 [-60.6 to -1.8]
  D6W3 between before/after lunch | -37.0 [-69.5 to -4.5] | -13.1 [-50.6 to 24.4]
  D7W3 between before/after lunch | -12.7 [-49.6 to 24.2] | -14.9 [-50.8 to 21.0]
  D8W3 between before/after lunch | -15.6 [-46.9 to 15.6] | -29.1 [-68.9 to 10.7]
  D2W3 between before/after evening meal | -37.8 [-75.3 to -0.3] | -15.6 [-45.1 to 13.8]
  D3W3 between before/after evening meal | -49.1 [-95.1 to -3.0] | -21.8 [-48.6 to 5.0]
  D4W3 between before/after evening meal | -42.6 [-86.1 to 0.8] | -24.2 [-49.5 to 1.1]
  D5W3 between before/after evening meal: number analyzed (Participants) | 13 | 13
  D5W3 between before/after evening meal | -31.5 [-70.7 to 7.6] | -5.2 [-39.1 to 28.7]
  D6W3 between before/after evening meal | -41.9 [-73.8 to -10.1] | -24.6 [-51.4 to 2.1]
  D7W3 between before/after evening meal | -33.6 [-72.7 to 5.4] | -4.4 [-36.6 to 27.9]
  D8W3 between before/after evening meal | -39.3 [-75.5 to -3.1] | -6.6 [-30.5 to 17.3]

15. Secondary Outcome: Change From Baseline in Mean Amplitude Glycemic Excursions (MAGE)
Description: Change from baseline in MAGE at each time points was calculated.
Time Frame: Baseline, up to 28 days
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Trelagliptin 100 mg | Alogliptin 25 mg
Number analyzed (Participants) | 13 | 14
mg/dL
  D2W3: number analyzed (Participants) | 13 | 13
  D2W3 | -28.42 [-50.55 to -6.29] | -47.25 [-77.78 to -16.71]
  D3W3: number analyzed (Participants) | 13 | 13
  D3W3 | -33.72 [-60.42 to -7.03] | -52.75 [-76.50 to -28.99]
  D4W3: number analyzed (Participants) | 13 | 13
  D4W3 | -36.08 [-64.14 to -8.03] | -44.67 [-69.51 to -19.83]
  D5W3: number analyzed (Participants) | 13 | 13
  D5W3 | -23.12 [-45.68 to -0.56] | -50.22 [-81.42 to -19.02]
  D6W3: number analyzed (Participants) | 13 | 13
  D6W3 | -38.05 [-67.39 to -8.70] | -34.82 [-62.54 to -7.09]
  D7W3: number analyzed (Participants) | 13 | 13
  D7W3 | -25.74 [-48.52 to -2.96] | -37.18 [-62.06 to -12.31]
  D8W3: number analyzed (Participants) | 13 | 13
  D8W3 | -24.26 [-44.71 to -3.82] | -41.38 [-66.75 to -16.01]

16. Secondary Outcome: Change From Baseline in Mean 24-hour Blood Glucose Levels
Description: Change from baseline in mean 24-hour blood glucose levels at each time points was calculated.
Time Frame: Baseline, up to 28 days
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Trelagliptin 100 mg | Alogliptin 25 mg
Number analyzed (Participants) | 13 | 14
mg/dL
  D2W3 | -8.14 [-20.37 to 4.09] | -16.77 [-23.33 to -10.21]
  D3W3 | -8.15 [-21.55 to 5.25] | -12.46 [-23.07 to -1.86]
  D4W3 | -13.12 [-23.02 to -3.21] | -15.85 [-23.57 to -8.13]
  D5W3 | -13.95 [-22.90 to -5.00] | -17.46 [-27.90 to -7.03]
  D6W3 | -8.37 [-17.30 to 0.56] | -15.79 [-24.43 to -7.14]
  D7W3 | -6.38 [-14.31 to 1.54] | -14.23 [-22.00 to -6.46]
  D8W3 | -8.46 [-21.29 to 4.37] | -14.94 [-21.97 to -7.90]

17. Secondary Outcome: Change From Baseline in Mean Daytime Blood Glucose Levels
Description: Change from baseline in mean daytime blood glucose levels at each time points was calculated.
Time Frame: Baseline, up to 28 days
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Trelagliptin 100 mg | Alogliptin 25 mg
Number analyzed (Participants) | 13 | 14
mg/dL
  D2W3 | -11.08 [-25.75 to 3.58] | -20.38 [-28.27 to -12.48]
  D3W3 | -12.48 [-26.87 to 1.91] | -17.21 [-29.46 to -4.97]
  D4W3 | -18.42 [-28.06 to -8.78] | -21.80 [-31.20 to -12.40]
  D5W3 | -19.53 [-29.75 to -9.31] | -22.54 [-35.28 to -9.81]
  D6W3 | -14.27 [-24.00 to -4.54] | -19.34 [-29.10 to -9.59]
  D7W3 | -10.86 [-20.48 to -1.25] | -16.92 [-26.10 to -7.75]
  D8W3 | -12.90 [-26.16 to 0.36] | -19.78 [-28.28 to -11.27]

18. Secondary Outcome: Change From Baseline in Mean Nocturnal Blood Glucose Levels
Description: Change from baseline in mean nocturnal blood glucose levels at each time points was calculated.
Time Frame: Baseline, up to 28 days
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Trelagliptin 100 mg | Alogliptin 25 mg
Number analyzed (Participants) | 13 | 14
mg/dL
  D2W3 | -2.65 [-17.20 to 11.89] | -10.69 [-23.02 to 1.64]
  D3W3 | 0.52 [-15.45 to 16.48] | -3.38 [-18.40 to 11.65]
  D4W3 | -3.17 [-18.50 to 12.16] | -3.76 [-15.40 to 7.89]
  D5W3 | -4.09 [-16.58 to 8.40] | -6.43 [-20.62 to 7.76]
  D6W3 | 5.55 [-6.57 to 17.68] | -7.98 [-20.46 to 4.51]
  D7W3 | 3.86 [-4.41 to 12.13] | -8.59 [-18.50 to 1.33]
  D8W3 | 1.06 [-13.04 to 15.16] | -5.96 [-17.16 to 5.24]

19. Secondary Outcome: Change From Baseline in AUC for Blood Glucose
Description: Change from baseline in AUC for blood glucose levels at each time points was calculated.
Time Frame: Baseline, up to 28 days
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: mg·min/dL
Arm/Group | Trelagliptin 100 mg | Alogliptin 25 mg
Number analyzed (Participants) | 13 | 14
mg·min/dL
  D2W3 | -2340.4 [-5859.6 to 1178.8] | -4828.9 [-6716.3 to -2941.6]
  D3W3 | -2348.4 [-6208.4 to 1511.6] | -3594.8 [-6648.1 to -541.5]
  D4W3 | -3723.2 [-6575.5 to -870.8] | -4565.6 [-6788.3 to -2343.0]
  D5W3 | -4017.8 [-6594.3 to -1441.4] | -5023.4 [-8025.0 to -2021.8]
  D6W3 | -2408.2 [-4978.6 to 162.3] | -4526.4 [-7012.3 to -2040.6]
  D7W3 | -1837.6 [-4117.9 to 442.7] | -4097.5 [-6332.3 to -1862.7]
  D8W3 | -2438.5 [-6134.2 to 1257.1] | -4302.9 [-6327.4 to -2278.5]

20. Secondary Outcome: Change From Baseline in AUC for Blood Glucose During Periods When Blood Glucose Levels Reached 110 mg/dL (Hypoglycemia)
Description: Change from baseline in AUC for blood glucose during periods when blood glucose levels reached 110 mg/dL at each time points was calculated.
Time Frame: Baseline, up to 28 days
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: mg·min/dL
Arm/Group | Trelagliptin 100 mg | Alogliptin 25 mg
Number analyzed (Participants) | 13 | 14
mg·min/dL
  D2W3 | -2263.8 [-5522.2 to 994.7] | -4735.1 [-6642.5 to -2827.7]
  D3W3 | -2479.2 [-6073.9 to 1115.4] | -3742.8 [-6840.0 to -645.5]
  D4W3 | -3755.3 [-6409.6 to -1101.0] | -4576.9 [-6710.1 to -2443.6]
  D5W3 | -3845.6 [-6396.3 to -1295.0] | -4812.0 [-7716.0 to -1908.0]
  D6W3 | -2581.9 [-4877.8 to -286.0] | -4592.1 [-7132.0 to -2052.3]
  D7W3 | -2184.1 [-4350.4 to -17.7] | -4169.3 [-6477.7 to -1860.8]
  D8W3 | -2634.2 [-5836.3 to 568.0] | -4335.7 [-6389.1 to -2282.4]

21. Secondary Outcome: Standard Deviation (SD) of 24-hour Blood Glucose Values
Time Frame: Baseline, up to 28 days
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Trelagliptin 100 mg | Alogliptin 25 mg
Number analyzed (Participants) | 13 | 14
mg/dL
  Baseline | 38.18 [27.46 to 48.91] | 40.44 [34.14 to 46.74]
  D2W3 | 30.68 [24.39 to 36.97] | 27.41 [22.11 to 32.71]
  D3W3 | 26.42 [22.32 to 30.53] | 25.20 [21.51 to 28.89]
  D4W3 | 26.48 [21.31 to 31.65] | 27.54 [23.69 to 31.39]
  D5W3 | 28.29 [23.82 to 32.77] | 27.16 [22.22 to 32.11]
  D6W3 | 25.44 [20.45 to 30.43] | 28.51 [23.13 to 33.89]
  D7W3 | 28.68 [24.10 to 33.27] | 29.54 [23.07 to 36.01]
  D8W3 | 30.84 [25.33 to 36.35] | 28.81 [23.37 to 34.26]

22. Secondary Outcome: Changes From Baseline in the SD of Daytime Blood Glucose Values
Description: Change from baseline in SD of daytime blood glucose values at each time points was calculated.
Time Frame: Baseline, up to 28 days
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Trelagliptin 100 mg | Alogliptin 25 mg
Number analyzed (Participants) | 13 | 14
mg/dL
  D2W3 | -9.78 [-19.01 to -0.54] | -13.28 [-21.07 to -5.48]
  D3W3 | -12.82 [-23.36 to -2.29] | -13.12 [-19.85 to -6.39]
  D4W3 | -11.98 [-22.91 to -1.04] | -10.98 [-16.68 to -5.28]
  D5W3 | -10.88 [-21.93 to 0.18] | -12.54 [-20.37 to -4.71]
  D6W3 | -11.94 [-21.55 to -2.33] | -10.44 [-19.45 to -1.43]
  D7W3 | -8.13 [-17.70 to 1.44] | -9.49 [-18.54 to -0.43]
  D8W3 | -6.49 [-14.98 to 2.00] | -10.81 [-18.56 to -3.07]

23. Secondary Outcome: Changes From Baseline in the SD of Nocturnal Blood Glucose Values
Description: Change from baseline in SD of nocturnal blood glucose values at each time points was calculated.
Time Frame: Baseline, up to 28 days
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Trelagliptin 100 mg | Alogliptin 25 mg
Number analyzed (Participants) | 13 | 14
mg/dL
  D2W3 | -0.71 [-7.36 to 5.95] | -2.45 [-13.78 to 8.88]
  D3W3 | -3.55 [-9.51 to 2.40] | -9.76 [-18.48 to -1.03]
  D4W3 | -4.06 [-13.05 to 4.92] | -7.86 [-18.87 to 3.14]
  D5W3 | -2.96 [-8.25 to 2.33] | -5.21 [-16.82 to 6.39]
  D6W3 | -5.67 [-12.26 to 0.93] | -8.23 [-17.41 to 0.95]
  D7W3 | -5.25 [-10.02 to -0.47] | -8.01 [-17.17 to 1.16]
  D8W3 | -2.93 [-9.26 to 3.40] | -6.64 [-14.48 to 1.20]

24. Secondary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events
Time Frame: Up to 29 days
Population: Safety Analysis Set (SAS), SAS was defined as participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Trelagliptin 100 mg | Alogliptin 25 mg
Number analyzed (Participants) | 13 | 14
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: Up to 29 days
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Alogliptin 25 mg | Trelagliptin 100 mg
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 1/13 | 2/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 25 mg (N=13) | Trelagliptin 100 mg (N=14)
Gastric mucosal lesion (Gastrointestinal disorders) | 0 | 1
Feeling abnormal (General disorders) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-02-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT02771093/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/93/NCT02771093/SAP_001.pdf